CLINICAL TRIAL: NCT05760807
Title: An Open Label Pilot Study of Intranasal Oxytocin for Methamphetamine Withdrawal in Women
Brief Title: Intranasal Oxytocin for Methamphetamine Withdrawal in Women
Acronym: mOXY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Turning Point (Other)
Collaborators: National Centre for Clinical Research on Emerging Drugs (NCCRED) (Unknown); Eastern Health (Other); Monash University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E21-014-75603; NCR3SF18 (Other Grant/Funding Number: NCCRED)
Record Dates: First submitted 2023-02-14; First posted 2023-03-08 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Methamphetamine Use Disorder
Keywords: Methamphetamine Use Disorder; Intranasal oxytocin; Actigraphy; Sleep

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intranasal oxytocin (Experimental): Participants will receive oxytocin by intranasal spray under clinician supervision (1 insufflation equating to an active dose of 24 IU) twice daily (i.e., 48 IU per day), delivered over 7 days of a residential inpatient withdrawal admission.
  Interventions: Drug: Oxytocin nasal spray

INTERVENTIONS:
Drug: Oxytocin nasal spray — Intranasal oxytocin, administered dose 24 international units (IU) twice daily, delivered over 7 days of a residential inpatient withdrawal admission.

SUMMARY:
Methamphetamine use disorder (MUD) is a significant public health concern with burden to individuals, families and health systems estimated to cost over $5 billion annually in Australia. In 2016/17 there were 49,670 Australian treatment episodes for MUD, the first step of which typically involves inpatient withdrawal. Currently there are no approved medications to help manage methamphetamine withdrawal and consequently many people drop out of treatment prematurely, leaving them vulnerable to relapse.

Oxytocin is a candidate medication that has the potential to increase treatment retention, reduce withdrawal syndrome severity, increase post-withdrawal treatment engagement and reduce relapse rates.

The aim of this pilot study is to investigate whether intranasal oxytocin can improve withdrawal treatment outcomes in adult women with MUD. The study will examine the feasibility of intranasal oxytocin as a treatment for methamphetamine withdrawal in women. This will be explored by assessing length of stay in residential withdrawal, withdrawal symptom severity, post-discharge treatment engagement and relapse rates in a group of women who are prescribed intranasal oxytocin during their medically supervised methamphetamine withdrawal at a residential detoxification program. The safety of intranasal oxytocin will also be assessed. A secondary objective of the study is to conduct an exploratory analysis regarding participants' capacity to interact effectively with others, as well as changes in social networks and/or engagement with therapeutic services.

There is an observational sub-study affiliated with this main pilot study that is optional for individuals recruited to the main pilot trial to additionally participate in. This sub-study aims to investigate how sleep quality and patterns change before, during, and after detoxification from methamphetamine in women. MUD and sleep disturbances have a complex bidirectional relationship. The use of methamphetamine is known to disrupt sleep quality and the circadian rhythm, although withdrawal from methamphetamine also induces significant sleep-wake cycle changes. There is evidence that methamphetamine disrupts functions regulated by the circadian rhythm. Furthermore, disruptions in circadian rhythms, including mutations in key genes, increases the propensity for addiction. Evaluation of how chronic methamphetamine use may disrupt rhythmicity, and vice versa, may provide invaluable information with regard to potential treatment options of methamphetamine use disorder. There has been little focus, so far, on the therapeutic potential of circadian rhythm modifiers as treatment options in the addiction space, as sleep disturbances have often been merely viewed as a consequence of substance use.

Specific to the sub-study, participants will be asked to wear an actigraphy watch. The actigraphy watch device will be worn for at least 7 days prior to, 7 days during, and 7 days post methamphetamine detoxification. This is the only difference between the sub-study and the main pilot study; there are no other additional requirements or assessments involved in the actigraphy sub-study.

ELIGIBILITY:
Inclusion Criteria:

* Adult females (sex assigned at birth) aged ≥18 to ≤65 years, admitted to the Turning Point Addiction Medicine Unit.
* Meeting DSM-5 criteria for Methamphetamine Use Disorder, moderate or severe (assessed by treating physician on pre-admission to residential withdrawal).
* Able to comply with study protocols.
* Able to provide informed consent to participate.

Exclusion Criteria:

* Non-English-speaking women.
* Women lactating, pregnant or of childbearing potential who are not willing to use an effective means of contraception for the duration of the trial.
* Meeting DSM-5 criteria for moderate-severe substance use disorder other than methamphetamine, nicotine and cannabis, as assessed by treating physician on pre-admission to residential withdrawal.
* Clinically significant or unmanaged medical or psychiatric illness (e.g., renal insufficiency, cirrhosis, unstable hypertension, unstable diabetes mellitus, seizure disorder, history of DSM-5 psychotic or bipolar disorder, current severe major depression, current suicidal ideation), assessed by treating physician on pre-admission to residential withdrawal.
* Current participation in another trial.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-03-29 (Actual); Primary Completion 2024-03-28 (Actual); Study Completion 2024-03-28 (Actual)

PRIMARY OUTCOMES:
Feasibility assessment | Screening to Admission Day 1
  Feasibility assessment, as measured by the proportion of screen failures compared to those who received the study drug.

SECONDARY OUTCOMES:
Length of stay in the inpatient withdrawal unit | Admission Day 1 to Admission Day 7
  Medical chart review to determine number of days stayed in the inpatient withdrawal unit.
Methamphetamine withdrawal symptom severity | Admission Day 1 to Admission Day 7
  Individual average score across the participants' length of stay in the inpatient withdrawal unit on the Amphetamine Withdrawal Questionnaire (scores on this measure range from 0 to 40 with higher score indicating greater severity).
Methamphetamine craving | Admission Day 1 to Admission Day 7
  Individual average score across the participants' length of stay in the inpatient withdrawal unit on the Visual Analogue Scale for Craving (scores on this measure range from 0 to 100, with higher scores indicating greater craving).
Sleep dysfunction | Admission Day 1 to Admission Day 7
  Individual average score across the participants' length of stay in the inpatient withdrawal unit on the Insomnia Severity Index (scores on this measure range from 0 to 28, with higher scores indicating greater sleep dysfunction).
Mood disturbance | Admission Day 1 to Admission Day 7
  Individual average score across the participants' length of stay in the inpatient withdrawal unit on the Abbreviated Profile of Mood States - Revised Version (total mood disturbance scores on this measure range from 0 to 116, with higher scores indicating greater disturbance)
Methamphetamine relapse | 1-month post-discharge
  Relapse is defined as a yes/no result for any methamphetamine use in the month following discharge from the withdrawal unit, as assessed using the Timeline Follow Back measure.
Treatment engagement | 1-month post-discharge
  Yes/No attendance at any form of treatment to assess treatment engagement at 1-month post-discharge.
Therapeutic alliance | 1-month post-discharge
  Working Alliance Inventory-Short Form Revised will be used to assess therapeutic alliance with nominated primary provider (scores on this measure range from 12 to 60, with higher scores indicating better therapeutic alliance).
Incidence of adverse events | Day 1 of admission to 1-month post-discharge
  Number and categorisation of reported adverse events.
Perceived burden of intranasal oxytocin | Admission Day 1 to Admission Day 7
  Individual average score across the participants' length of stay in the inpatient withdrawal unit on the Visual Analogue Scale for Medication Utilisation Burden (scores on this measure range from 0 to 100, with higher scores indicating greater perceived burden).
Perceived satisfaction with intranasal oxytocin | Admission Day 3 and 7
  Satisfaction with medication based on results from the Treatment Satisfaction Questionnaire (scores on this measure range from 0 to 100, with higher scores indicating greater satisfaction).
Severity of Clinical Condition | Baseline to 1-month post-discharge
  Change in clinician-rated assessment of the participant's condition using the Clinical Global Impression - Severity Scale (scores on this measure range from 1 to 7, with higher scores indicating poorer condition).
Improvement of Clinical Condition | 1-month post-discharge
  Clinician-rated assessment of the participant's overall clinical condition, substance use, and related problems compared to a baseline assessment, using the Clinical Global Impression - Improvement Scale (scores on this measure range from 5 to 35, with higher scores indicating a worsening of condition in comparison to baseline).

OTHER OUTCOMES:
Change in facial emotion recognition | Baseline to 1-month post-discharge
  Change in total score on the Facial Emotion Recognition Task at 1-month post-discharge compared to baseline.
Change in mentalisation | Baseline to 1-month post-discharge
  Change in total score on the Reading the Eyes in the Mind Task at 1-month post-discharge compared to baseline.
Change in social functioning | Baseline to 1-month post-discharge
  Change in score on the Social Functioning Scale at 1-month post-discharge compared to baseline (scores on this measure range from 0 to 24, with higher scores indicating poorer social functioning).
Sleep-wake cycles [part of the optional sub-study] | 7 days prior to, 7 days during, and 7 days post methamphetamine detoxification.
  Change in sleep-wake cycles, as assessed via actigraphy monitoring, before, during and after methamphetamine detoxification.
Objective assessment of sleep quality [part of the optional sub-study] | 7 days prior to, 7 days during, and 7 days post methamphetamine detoxification.
  Change in sleep quality, as assessed via actigraphy monitoring, before, during and after methamphetamine detoxification.
Objective assessment of sleep duration [part of the optional sub-study] | 7 days prior to, 7 days during, and 7 days post methamphetamine detoxification.
  Change in sleep duration, as assessed via actigraphy monitoring, before, during and after methamphetamine detoxification.
Subjective sleep quality | Baseline to 1-month post-discharge.
  Change in score on the Pittsburgh Sleep Quality Index at 1-month post-discharge compared to baseline (scores on this measure range from 0 to 21, with higher scores indicating poorer sleep quality).
Rhythmicity of sleep-wake cycles | Baseline to 1-month post-discharge.
  Sleep rhythmicity and categorisation of morning-evening preference grouping using the Morningness-Eveningness Questionnaire-Reduced Scale (scores on this measure range from 4-25, where higher scores are indicative of morning-type preferences - scores are categorised into one of 5 preference groups, ranging from "Definitely Evening Type" to "Definitely Morning Type").

CONTACTS AND LOCATIONS:
Overall Officials: Shalini Arunogiri, Principal Investigator — Turning Point, Eastern Health, Monash University
Locations (1):
- Turning Point, Richmond, Victoria, Australia